CLINICAL TRIAL: NCT02304029
Title: Usefulness of Sodium MRI in the Presurgical Assessment of Drug-resistant Partial Epilepsy
Acronym: EPISODIUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-27
Record Dates: First submitted 2014-11-20; First posted 2014-12-01 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Epileptic Seizures
Keywords: epilepsy; seizures
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- assessment of a innovative MRI (Experimental): Sodium MRI will be performed at CEMEREM, CHU Timone, the only site with this technique, with a Siemens Verio 3T MRI using a dedicated coil and a sequence already developed locally, in 90 patients with partial drug -resistant epilepsy
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI

SUMMARY:
Epilepsy is a common disease affecting 0.5 to 1% of the general population. Epilepsies refractory to drug treatment lead to increased morbidity, mortality and high costs for public health (representing 75% of the costs associated with epilepsy is among the most costly diseases in Neurology). The only curative therapy is surgical removal or disconnection of the epileptogenic network. To do this, a comprehensive presurgical evaluation is essential to accurately define the location of the epileptogenic zone (EZ) and its relationship with the functional areas that must be preserved. This approach requires in some cases intracerebral EEG recordings. This latter technique, expensive and invasive, remains at present, the standard method in the location of the ZE. In this context, the development of non-invasive and inexpensive methods is a priority in the field. Moreover, many fundamental studies have shown changes in ion homeostasis including sodium associated with hyperexcitability related to epilepsy. The investigators team at CEMEREM, CHU Timone, specialized in the development and validation of innovative methods in MRI, has developed an in vivo sodium MRI acquisition and processing of data unique in France, capable of quantifying the intracerebral sodium concentration in three dimensions in a completely non-invasive and non-irradiating manner

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a drug-resistant partial epilepsy for which an indication is indicated after préchirugical balance assessment.
* Patient not presenting a psychiatric disease chronicles, an demential syndrome,
* Patient not presenting contraindication to the realization of an examination by MRI

Exclusion Criteria:

* Patient suffering a not operable shape of partial epilepsy or a generalized epilepsy
* Patient suffering an evolutionary associated serious illness (cancer, autoimmune disease, hepatic insufficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Interest of Sodium MRI in the management of patients for localizing the EZ responsible for seizures that must be removed surgically to cure patients | 3 years
  The location of significant abnormal sodium concentrations will be compared to the location of surgical excision and faced with post-surgical results. The number of concordant and discordant locations (locations of sodium concentration abnormalities/ surgical cavity) It will be allowed the sensitivity, specificity, positive predictive value and negative predictive value of our technique ( patients free of seizures compare non-free patients crises postoperatively)

SECONDARY OUTCOMES:
etablish links between brain ionic changes and brain abnorman electrical activities | 3years
  Comparing the location of sodium abnormalities with the location of electrical abnormalities recorded in surface (EEG) or depth (SEEG) will allow us to establish links between ionic changes and abnormal electrical activity

CONTACTS AND LOCATIONS:
Overall Officials: Maxime GUYE, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (4):
- France (4):
  - Assistance Publique - Hopitaux de Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU NICE, Nice
  - CHU Nimes, Nîmes